CLINICAL TRIAL: NCT05365152
Title: The Effects of Partial Calories Replacement Using Substitute Meals on Glycemic Control During Short-term Insulin Intensive Therapy in Patients With Type 2 Diabetes
Brief Title: The Effect of Meal Replacement on the Time to Reach the Blood Glucose Target in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-793
Record Dates: First submitted 2022-04-14; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; Blood Sugar; High
Keywords: type 2 diabetes; Meal Replacement
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal replacement intervention group (Experimental): On the day of the patient's admission, the total calories required for the diabetic diet during the hospitalization period were calculated according to "ideal weight * 25/kcal" (BMI > 28, 80% of this value). Carbohydrates, fats, and proteins accounted for 50%, 30%, and 20% of the energy supply, respectively, and the calories of the three meals were distributed according to 1:2:2. The meal replacement intervention group replaced the daily meal with meal replacement on the basis of the conventional diabetic diet. About 400kcal calories in carbohydrates.
  Interventions: Dietary Supplement: Meal Replacement
- diabetes diet group (No Intervention): On the day of the patient's admission, the total calories required for the diabetic diet during the hospitalization period were calculated according to "ideal weight * 25/kcal" (BMI > 28, 80% of this value). Carbohydrates, fats, and proteins accounted for 50%, 30%, and 20% of the energy supply, respectively, and the calories of the three meals were distributed according to 1:2:2.

INTERVENTIONS:
Dietary Supplement: Meal Replacement — Meal Replacement
  Arms: Meal replacement intervention group

SUMMARY:
This study was designed as a randomized controlled study. It was planned to include 100 patients with type 2 diabetes who received short-term intensive insulin therapy and randomly divided them into a meal replacement intervention group and a conventional diabetes diet group according to 1:1. Both groups were treated with short-term intensive insulin therapy to control blood sugar. .

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients who meet the diagnosis of type 2 diabetes (CDS2020) and are willing to receive intensive insulin hypoglycemic therapy;
2. Glycated hemoglobin A1c≥7.5%;
3. Age between 18-70 years old, body mass index (BMI) 20-35kg/m2;
4. Be able and willing to cooperate with diet and exercise and monitor blood sugar in accordance with the project regulations, and agree to sign the informed consent.

Exclusion Criteria:

1. Diagnosed as type 1 diabetes or special type of diabetes;
2. Allergic or intolerable to the meal replacement food used in the study;
3. Acute complications of diabetes (including DKA, HHS, lactic acidosis)
4. Severe microvascular complications: proliferative retinopathy; urine AER>300mg/g or urine protein positive, quantitative>0.5g/d; uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy;
5. Significant macrovascular complications: patients with acute cerebrovascular accident, acute coronary syndrome, peripheral arterial disease requiring vascular intervention or amputation within 12 months before enrollment;
6. Serum creatinine clearance rate is less than 50ml/min/1.73m2 (calculated according to CKDEPI formula), alanine aminotransferase ≥ 3 times the upper limit of normal, and total bilirubin ≥ 2 times the upper limit of normal;
7. The cumulative time of using drugs that may affect blood sugar for more than 1 week within 12 weeks, such as oral/intravenous glucocorticoids, GH, estrogen/progestin, high-dose diuretics, antipsychotics, etc.;
8. Systemic infection or serious concomitant diseases; patients with malignant tumors or chronic diarrhea;
9. Uncontrolled endocrine gland dysfunction;
10. Mental or communication disorders;
11. Pregnant and lactating women;
12. The subject is not cooperative, or the investigator judges that it may be difficult to complete the investigator;
13. Other circumstances judged by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time required for blood sugar to reach target | 7-10days
  The time it takes for the patient to reach the prescribed glycemic control goals during the hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No